CLINICAL TRIAL: NCT03991429
Title: Higher Neural Contribution Underlying Lower Urinary Tract Symptoms in Men With Benign Prostatic Hyperplasia Undergoing Bladder Outlet Procedures.
Brief Title: Brain Imaging in Men With Lower Urinary Tract Symptoms
Status: Completed | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Rose Khavari, M.D., Principal Investigator, Houston Methodist Hospital Urologist & Research Director, The Methodist Hospital Research Institute
Other Study IDs: Pro00020695
Record Dates: First submitted 2019-01-02; First posted 2019-06-19 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Voiding Disorders
Keywords: Voiding dysfunction; Benign Prostatic Hyperplasia (BPH); Lower urinary tract symptoms (LUTS); Functional Magnetic Resonance Imaging; Urodynamic studies
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Urodynamics; Surveys and Questionnaires; Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with BPH and significant improvement in storage symptoms after BOO procedures
  Interventions: Diagnostic Test: Simultaneous functional MRI and urodynamic studies; Behavioral: Questionnaires; Other: Post Void Residual (PVR), Uroflow and Bladder Diary; Diagnostic Test: Urinalysis
- Group 2: Patients with BPH who have persistent storage symptoms after BOO procedures
  Interventions: Diagnostic Test: Simultaneous functional MRI and urodynamic studies; Behavioral: Questionnaires; Other: Post Void Residual (PVR), Uroflow and Bladder Diary; Diagnostic Test: Urinalysis
- Group 3 (Control group): Men without LUTS who are planning to undergo radical prostatectomy
  Interventions: Diagnostic Test: Simultaneous functional MRI and urodynamic studies; Behavioral: Questionnaires; Other: Post Void Residual (PVR), Uroflow and Bladder Diary; Diagnostic Test: Urinalysis

INTERVENTIONS:
Diagnostic Test: Simultaneous functional MRI and urodynamic studies — Double lumen 7 Fr MRI-compatible catheters will be placed in the bladder and rectum. A Phillips Ingenia 3.0T full body MRI scanner with standard 12 channel head coil will be used. Instructions to communicate using right hand signals representing "full urge" and "voiding or attempt of voiding" will be given. Signs will be shown to the patient when filling of the bladder is begun and when filling is stopped. Also, in order to keep our noise-to-signal ratio low, all stimulators including any extra visual stimuli and the UDS machine will be removed from the MRI scanner room. The filling and voiding cycle will be repeated up to 4 times in each patient. Bladder will be aspirated after each voiding. This algorithm will be performed before, and, 3 and 6 months following BOO procedure.
Behavioral: Questionnaires — Each patient will provide a detailed history and undergo a complete physical examination. Each patient will have the following assessments: IPSS and Incontinence Severity Index (ISI), Patient Global impression of severity (PGI-S) and improvement (PGI-I), International Index of Erectile Function (IIEF-5), MRI Safety Screening Questionnaire.
Other: Post Void Residual (PVR), Uroflow and Bladder Diary — Follow-up assessments: Uroflow and PVR assessment, bladder diary, and all questionnaires will be repeated in all patients at one, three, and six months.
Diagnostic Test: Urinalysis — Urine sample

SUMMARY:
Benign Prostatic Hyperplasia (BPH) affects the storage and voiding phases of the micturition cycle. Lower urinary tract symptoms (LUTS) refers to storage symptoms such as urinary frequency, urgency, urge urinary incontinence and nocturia. Surgical options for bladder outlet obstruction (BOO), including prostate ablation and transurethral resection, are currently offered for symptomatic improvement. However, 30% of patients report persistent LUTS after BOO procedures. Neuroplasticity induced by BPH and BOO can be contributory of persistent LUTS in these men, having different brain activation patterns during the micturition cycle. The investigators proposed unique multimodal functional Magnetic Resonance Imaging (fMRI) study that will identify for the first time, structural and functional brain contributions to LUTS in men with BPH and BOO at baseline and following BOO procedures. The investigators hypothesize that men with symptomatic BPH who have persistent LUTS following BOO procedures have a distinct brain activation pattern in Regions of Interest (RoI) that regulate the micturition cycle.

DETAILED DESCRIPTION:
The investigators propose a unique, multimodal prospective study that will allow investigators to identify for the first time the structural and functional brain contributions to LUTS in men with BPH and BOO at baseline and post procedure. For this, The investigators will recruit three different groups of patients:

Group 1: Patients with BPH and significant improvement in the storage symptoms following BOO procedures.

Group 2: Patients with BPH who have persistent storage symptoms following BOO procedures.

Group 3 (CONTROL GROUP): Men without LUTS who are planning to undergo radical prostatectomy.

Each participant will provide a detailed history, undergo a complete physical examination and will have the following assessments: IPSS, IPSS Quality of life, Incontinence Severity Index (ISI), Patient Global impression of severity (PGI-S) and improvement (PGI-I)19, 20, International Index of Erectile Function (IIEF-5), MRI Safety Screening Questionnaire. A post void residual volume will be measured and a urine sample will be obtained for urinalysis (patients and controls). A two-day bladder diary will also be obtained from the participants. Participants in group 1 and 2 will undergo a clinical urodynamic study within a year prior to the neuroimaging scan. All participants will be followed up at one, three and six months after the BOO procedures (Transurethral resection/ablation of prostate and simple prostatectomy) and radical prostatectomy in the control group. On each visit, the investigators will gather the following data: Uroflow and PVR assessment, bladder diary, and all questionnaires will be repeated in all patients at one, three, and six months. Participants with persistent storage LUTS at six months will have a repeat UDS to ensure BOO is resolved. Group 1 and 2 will undergo simultaneous fMRI/UDS scanning twice during this study: First before BOO procedures and at the second one at six months. The control group will undergo baseline fMRI/UDS.

Investigators' established platform for simultaneous urodynamic study and functional MRI scanning will allow investigators to detect structural changes during the micturition cycle. Providing 3D structural images and functional images to have a better understanding of the brain effect on LUTS. By correlating the bold signal changes, structural markers and participant's clinical data, investigators will provide scientific rationale for subsequent studies in the field of neurourology.

ELIGIBILITY:
Inclusion Criteria:

* Controls (n=13) Men older than 45 years undergoing radical prostatectomy without LUTS
* IPSS (International prostate symptom score lower than 12)
* Nocturia equal or less than 2 on a two day bladder diary
* Group 1 (n=18) Men older than 45 with improved LUTS after 6 months of a BOO procedure and IPSS less than 12
* Improvement in IPSS in at least 3 points for storage symptoms
* Nocturia equal or less than 2 on a two day bladder diary
* Group 2 (n=9) Men older than 45 with persistent LUTS at six months post BOO procedure
* IPSS higher than 8
* Nocturia more than 2
* Delta change in IPSS score less than negative 3 points

Exclusion Criteria:

* Men with
* Neurogenic bladder
* Urethral stricture
* Prior BOO procedures
* History of urinary retention with indwelling foley catheter or intermittent catheterization Additional exclusion criteria for Group 1 and 2 (Subjects with BPH and LUTS)
* History of bladder cancer within 5 years
* History of treatment for prostate cancer other than active surveillance
* Intradetrusor injection of BTX-A within 9 months prior to screening for any urological condition

Ages: 45 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with benign prostatic hyperplasia
Study Population: Houston Methodist Hospital has four fulltime fellowship-trained Urologists in the field of functional Urology and voiding dysfunction who perform over 300 Bladder Outlet Obstruction procedures per year. Patients for our study will be recruited from our clinics
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Blood Oxygen Level Dependent (BOLD) signals | 1 year
  BOLD signal intensity in the Regions of Interest at the point of "full urge" at baseline and following Bladder Outlet Obstruction (BOO) procedures in groups 1, 2, and controls.

SECONDARY OUTCOMES:
Fractional Anisotropy (FA) | 1 year
  FA; Fractional anisotropy (FA) is a scalar value between zero and one that describes the degree of anisotropy of a diffusion process. A value of zero means that diffusion is isotropic, i.e. it is unrestricted (or equally restricted) in all directions. No units.
Mean Diffusivity (MD) | 1 year
  Mean diffusivity of Anterior Thalamic Radiation (ATR) and Superior Longitudinal Fasciculus (SLF) white matter tracts in groups 1,2, and controls. MD is a scalar value between zero and one that describes the degree of diffusivity. No units.
Uroflow measure | 1 year
  Maximum Qmax of urine (ml/sec): The range is between 0-40 ml/ sec.
Postvoid Residual | 1 year
  Postvoid Residual (PVR) of urine in mL: The range is between 0-900 ml.
Urinary symptoms scores | 1 year
  Urinary symptoms scores (no unit): The range is between 0-35

CONTACTS AND LOCATIONS:
Overall Officials: Rose Khavari, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States